CLINICAL TRIAL: NCT03285087
Title: Risk Prediction and Consequences of Dexmedetomidine-associated Hemodynamic Instability in Intubated Mechanically Ventilated Intensive Care Unit Patients
Brief Title: Risk Prediction of Dexmedetomidine-associated Hemodynamic Instability
Acronym: DEXSEDATION
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: dexmedetomidine is unavailable in this time
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200062
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The primary end point will be the occurrence of at least 1 episode of clinically significant hemodynamic instability during dexmedetomidine therapy defined as systolic blood pressure (SBP) < 80 mm Hg, diastolic blood pressure (DBP) <50 mm Hg, or heart rate <50 beats per minute (bpm) To qualify as an event, the hemodynamic variable had to remain below the specified threshold for at least 2 consecutive readings (≥30 minutes of recorded hemodynamic instability). The cumulative incidence of hemodynamic instability events during dexmedetomidine sedation will be plotted and Cox proportional hazards models will be constructed to determine hazard ratios (HRs) and 95% confidence intervals (CIs) for the risk factors of hemodynamic instability during dexmedetomidine therapy.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEX 0.2 μg/kg/h (Experimental): Patients will receive dexmedetomidine for sedation with initial maintenance dose rate of 0.2 μg/kg/h. The dose will be increased in 0.1 μg/kg/h increments to achieve target Richmond Agitation Sedation Scale (RASS) levels of -2 to zero and with a maximum dose of 1.4 μg/kg/h for 24 hours.
  Interventions: Drug: DEX 0.2 μg/kg/h.

INTERVENTIONS:
Drug: DEX 0.2 μg/kg/h. — DEX 0.2 μg/kg/h. The dose will be increased in 0.1 μg/kg/h increments to achieve target Richmond Agitation Sedation Scale (RASS) levels of -2 to zero and with a maximum dose of 1.4 μg/kg/h for 24 hours.
  Other Names: Precedex

SUMMARY:
Hypotension and bradycardia have been commonly associated with dexmedetomidine therapy, occurring in 13% to 68% and 1% to 42% of patients, respectively. The variability in reported incidence may be partially attributed to inconsistent definitions and study populations. The significance of this hemodynamic instability is not only highlighted by its high incidence but also the need for corrective interventions. In one study, hemodynamic instability requiring clinical intervention occurred in nearly one third of ICU patients receiving dexmedetomidine. Moreover, patients who experienced dexmedetomidine-associated hypotension had a higher mortality rate than those who did not.

DETAILED DESCRIPTION:
Dexmedetomidine is specific for the α-2a receptor, especially at lower concentrations, resulting in both vasodilation and a blunting of the sympathetic response. Due to these mechanistic considerations, patients who are dependent upon adrenergic tone to maintain blood pressure are more prone to its' hemodynamic instability. This is especially true in those who are receiving dexmedetomidine in the settings of hypovolemia, traumatic spinal cord injury, or general anesthetic administration. The use of dexmedetomidine in these patient populations may explain the high rate of hypotension reported in a recent study in trauma patients where almost 50% of patients had a spinal cord injury.

Although hemodynamic instability may negatively impact outcomes in the ICU, specific risk factors for the development of clinically significant hemodynamic instability in patients receiving dexmedetomidine are poorly characterized in the current literature. Although previous studies in focused populations have implicated dexmedetomidine dosing strategies, including initial loading infusions and titration frequency, the degree to which alternative patient-specific factors or concurrent interventions impact the risk of hemodynamic instability remains incompletely understood.

The aim of this study will be to determine the risk factors of dexmedetomidine-associated hemodynamic instability in critically ill trauma patients and the effect of this hemodynamic instability on different body systems.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years old)
* admitted to Intensive care units in Assiut university Hospital
* requiring endotracheal intubation, mechanical ventilation and light to moderate sedation
* of an estimated duration not less than 24h.

Exclusion Criteria:

* History of coronary care unit admission.
* Severe traumatic brain injury.
* Low baseline arterial blood pressure defined as SBP <100 mm Hg or mean arterial blood pressure (MAP) <70 mm Hg in the 60 minutes preceding dexmedetomidine initiation.
* Slow baseline heart rate was <70 bpm in the 60 minutes preceding dexmedetomidine initiation.
* Spinal cord injury.
* Patients who have a cardiac pacemaker or automatic implantable cardioverter defibrillator.
* Patients who are admitted with a primary diagnosis of substance withdrawal.
* Pregnant females.
* Patients who are incarcerated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of hemodynamic instability events during dexmedetomidine | 24 hours
  The primary end point will be the occurrence of at least 1 episode of clinically significant hemodynamic instability during dexmedetomidine therapy defined as systolic blood pressure (SBP) < 80 mm Hg, diastolic blood pressure (DBP) <50 mm Hg, or heart rate <50 beats per minute (bpm) To qualify as an event, the hemodynamic variable had to remain below the specified threshold for at least 2 consecutive readings (≥30 minutes of recorded hemodynamic instability). The cumulative incidence of hemodynamic instability events during dexmedetomidine sedation will be plotted and Cox proportional hazards models will be constructed to determine hazard ratios (HRs) and 95% confidence intervals (CIs) for the risk factors of hemodynamic instability during dexmedetomidine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor of anesthesia, faculty of medicine, Assiut university, Egypt; Hala S Abdelghaffar, MD, Principal Investigator — Professor of anesthesia, faculty of medicine, Assiut university, Assiut, Egypy
Locations (1):
- Assiut university main hospital, Trauma ICU, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No